CLINICAL TRIAL: NCT00712036
Title: Entry Into Comprehensive Methadone Treatment Via Interim Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA R01 13636; R01DA013636 (NIH)
Record Dates: First submitted 2008-07-02; First posted 2008-07-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Opiate Dependence
Keywords: Heroin dependence; Interim Methadone Treatment; Counseling
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — Denture, Partial, Temporary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interim (Active Comparator): Methadone maintenance for up to 4 months with emergency counseling only for individuals on program waiting lists.
  Interventions: Behavioral: Interim
- Comprehensive (Active Comparator): Methadone Treatment provided with counseling as usual.
  Interventions: Behavioral: Comprehensive
- Restored (Active Comparator): Methadone Treatment with counseling provided by a clinician with a lower caseload than counseling as usual.
  Interventions: Behavioral: Restored

INTERVENTIONS:
Behavioral: Interim — Methadone maintenance with emergency counseling only for up to 4 months
  Arms: Interim
Behavioral: Comprehensive — Methadone treatment with counseling as usual
  Arms: Comprehensive
Behavioral: Restored — Methadone maintenance with counseling provided by a clinician with a lower than usual caseload
  Arms: Restored

SUMMARY:
The purpose of the study is to determine whether one of three levels of counseling intensity will be associated with better treatment outcomes when combined with methadone maintenance treatment for heroin-addicted adults drawn from a methadone treatment program waiting list.

DETAILED DESCRIPTION:
Waiting lists for methadone treatment programs persist, and new and more effective approaches for expanding treatment access and improving outcomes for heroin dependent individuals are needed. Recently completed research demonstrated that so-called "Interim Methadone Maintenance" (i.e., methadone with crisis counseling only, for individuals on waiting lists) was associated with greater entry into methadone treatment, less self-reported heroin and cocaine use, lower rates of opioid-positive drug tests, and lower rates of self-reported crime. The present study will build on this work by comparing three levels of counseling provided with methadone treatment: 1)"Interim" Methadone Treatment; 2) "Comprehensive" Methadone Treatment (which is the name for the usual amount of counseling provided, i.e., about once per week) and; 3)"Restored" Methadone Treatment in which the counselors will have a lower case load and will be able to provide more attention to their patients.

ELIGIBILITY:
Inclusion Criteria:

* adult
* meets criteria for methadone maintenance
* unable to gain admission to methadone program within 14 days

Exclusion Criteria:

* pregnant
* acute medical or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Opioid positive drug tests | 4 and 12 months post-baseline

SECONDARY OUTCOMES:
HIV risk behavior | 4 and 12 months post-baseline
Treatment Retention | 4 and 12 months post-baselin
Cost-benefit | 12 months post-baseline
Cocaine positive tests | 4 and 12 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Schwartz RP, Jaffe JH, Highfield DA, Callaman JM, O'Grady KE. A randomized controlled trial of interim methadone maintenance: 10-Month follow-up. Drug Alcohol Depend. 2007 Jan 5;86(1):30-6. doi: 10.1016/j.drugalcdep.2006.04.017. Epub 2006 Jun 21. PMID 16793221
- [Background] Schwartz RP, Highfield DA, Jaffe JH, Brady JV, Butler CB, Rouse CO, Callaman JM, O'Grady KE, Battjes RJ. A randomized controlled trial of interim methadone maintenance. Arch Gen Psychiatry. 2006 Jan;63(1):102-9. doi: 10.1001/archpsyc.63.1.102. PMID 16389204
- [Background] Highfield DA, Schwartz RP, Jaffe JH, O'Grady KE. Intravenous and intranasal heroin-dependent treatment-seekers: characteristics and treatment outcome. Addiction. 2007 Nov;102(11):1816-23. doi: 10.1111/j.1360-0443.2007.01998.x. Epub 2007 Sep 3. PMID 17784892
- [Background] Schwartz RP, Kelly SM, O'Grady KE, Gandhi D, Jaffe JH. Interim methadone treatment compared to standard methadone treatment: 4-month findings. J Subst Abuse Treat. 2011 Jul;41(1):21-9. doi: 10.1016/j.jsat.2011.01.008. Epub 2011 Feb 24. PMID 21353445
- [Result] Schwartz RP, Alexandre PK, Kelly SM, O'Grady KE, Gryczynski J, Jaffe JH. Interim versus standard methadone treatment: a benefit-cost analysis. J Subst Abuse Treat. 2014 Mar;46(3):306-14. doi: 10.1016/j.jsat.2013.10.003. Epub 2013 Oct 14. PMID 24239030
- [Result] Schwartz RP, Kelly SM, O'Grady KE, Gandhi D, Jaffe JH. Randomized trial of standard methadone treatment compared to initiating methadone without counseling: 12-month findings. Addiction. 2012 May;107(5):943-52. doi: 10.1111/j.1360-0443.2011.03700.x. Epub 2012 Feb 11. PMID 22029398
- [Result] Kelly SM, Schwartz RP, O'grady KE, Gandhi D, Jaffe JH. Impact of methadone with versus without drug abuse counseling on HIV risk: 4- and 12-month findings from a clinical trial. J Addict Med. 2012 Jun;6(2):145-52. doi: 10.1097/ADM.0b013e31823ae556. PMID 22134175